CLINICAL TRIAL: NCT06169735
Title: Does Fluorescence With or Without Indocyanine Green Improve Parathyroid Identification and Preservation
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Stryker Nordic (Industry)
Responsible Party: Principal Investigator, Herbert Chen, Professor, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-300011872; Stryker (Other: Stryker)
Record Dates: First submitted 2023-12-05; First posted 2023-12-13 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Parathyroid Dysfunction; Adenoma
Keywords: Indocyanine Green; Parathyroid Surgery
MeSH Terms: conditions — Parathyroid Diseases; Adenoma | interventions — Indocyanine Green

STUDY DESIGN:
Intervention Model Description: This is already a pre-approved drug by FDA.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Parathyroid patients (Experimental): patients who require parathyroid identification and preservation during parathyroid surgery maneuver
  Interventions: Drug: Indocyanine green; Device: SPY Portable Handheld Imaging

INTERVENTIONS:
Drug: Indocyanine green — ICG Administration: All enrolled patients with scheduled thyroidectomy or parathyroidectomy will receive a standard cervical incision that afford access to either side of neck. Following sufficient exposure of thyroid, 25 mg of indocyanine green (ICG), reconstituted in 10 ml of sterile water, will be administered intravenously. A dosage of 1 ml of this solution will be injected into a peripheral IV line, followed by a 5 ml flush of normal saline to ensure the propagation of the dye within the vascular compartment.
Device: SPY Portable Handheld Imaging — Fluorescent Imaging: Approximately 30 seconds post-administration, the parathyroid glands are expected to exhibit fluorescence under near-infrared imaging. The emitted fluorescence is anticipated to persist for approximately 20 minutes, allowing ample time for intraoperative evaluation of parathyroid viability and perfusion
  Other Names: SPY-PHI

SUMMARY:
The aim of this study is to determine if fluorescence with or without indocyanine green can facilitate safe and accurate thyroid and parathyroid surgery.

DETAILED DESCRIPTION:
The accurate identification of the parathyroid gland is a crucial aspect of thyroid and parathyroid surgery. Failing to recognize the parathyroid gland during thyroidectomy can result in the inadvertent removal of the gland, leading to postoperative hypocalcemia. On the other hand, during parathyroidectomy, there is a risk of mistaking other structures, such as lymph nodes, for parathyroid adenomas, which can leave the patient without a cure. Currently UAB employs intraoperative PTH or radioactive isotope techniques in conjunction with surgeon judgment. However, both methods have limitations, including being time-consuming, posing logistical challenges, and not providing feedback before gland removal.

Parathyroid fluorescence is a relatively new technology. It was initially discovered that the parathyroid gland emits fluorescence, which distinguishes it from the surrounding tissues. Additionally, indocyanine green dye is readily taken up by the parathyroid gland, making its detection easy to the naked eye. Research has demonstrated that parathyroid fluorescence, with or without indocyanine green, is not only safe but also helps reduce postoperative hypocalcemia and locate lesions in patients with imaging-negative parathyroid adenomas. However, the current use of parathyroid fluorescence is not standardized, and further studies are needed to explore its clinical utility in terms of cure rates and postoperative complications.

ELIGIBILITY:
Inclusion Criteria:

* age greater than 18 years old

Exclusion Criteria:

* Patients with iodine or shellfish allergies would be excluded.
* Patients with allergy to indocyanine green.
* Pregnancy

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 417 (Estimated)
Dates: Start 2024-04-11 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of Parathyroid Glands identified by ICG | 20 minutes
  Measuring the percentage of the number of glands per participant that emit fluorescence.
  ICG Administration: All enrolled patients with scheduled thyroidectomy or parathyroidectomy will receive a standard cervical incision that afford access to either side of neck. Following sufficient exposure of thyroid, 25 mg of indocyanine green (ICG), reconstituted in 10 ml of sterile water, will be administered intravenously. A dosage of 1 ml of this solution will be injected into a peripheral IV line, followed by a 5 ml flush of normal saline to ensure the propagation of the dye within the vascular compartment.
  Fluorescent Imaging: Approximately 30 seconds post-administration, the parathyroid glands are expected to exhibit fluorescence under near-infrared imaging. The emitted fluorescence is anticipated to persist for approximately 20 minutes, allowing ample time for intraoperative evaluation of parathyroid viability and perfusion.

CONTACTS AND LOCATIONS:
Overall Officials: Herbert Chen, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB Callahan Eye, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Edafe O, Antakia R, Laskar N, Uttley L, Balasubramanian SP. Systematic review and meta-analysis of predictors of post-thyroidectomy hypocalcaemia. Br J Surg. 2014 Mar;101(4):307-20. doi: 10.1002/bjs.9384. Epub 2014 Jan 9. PMID 24402815
- [Background] Carter Y, Chen H, Sippel RS. An intact parathyroid hormone-based protocol for the prevention and treatment of symptomatic hypocalcemia after thyroidectomy. J Surg Res. 2014 Jan;186(1):23-8. doi: 10.1016/j.jss.2013.09.026. Epub 2013 Oct 8. PMID 24144426
- [Background] Desiato V, Melis M, Amato B, Bianco T, Rocca A, Amato M, Quarto G, Benassai G. Minimally invasive radioguided parathyroid surgery: A literature review. Int J Surg. 2016 Apr;28 Suppl 1:S84-93. doi: 10.1016/j.ijsu.2015.12.037. Epub 2015 Dec 23. PMID 26721192
- [Background] Noureldine SI, Gooi Z, Tufano RP. Minimally invasive parathyroid surgery. Gland Surg. 2015 Oct;4(5):410-9. doi: 10.3978/j.issn.2227-684X.2015.03.07. PMID 26425454
- [Background] Paras C, Keller M, White L, Phay J, Mahadevan-Jansen A. Near-infrared autofluorescence for the detection of parathyroid glands. J Biomed Opt. 2011 Jun;16(6):067012. doi: 10.1117/1.3583571. PMID 21721833
- [Background] Silver Karcioglu AL, Triponez F, Solorzano CC, Iwata AJ, Abdelhamid Ahmed AH, Almquist M, Angelos P, Benmiloud F, Berber E, Bergenfelz A, Cha J, Colaianni CA, Davies L, Duh QY, Hartl D, Kandil E, Kim WW, Kopp PA, Liddy W, Mahadevan-Jansen A, Lee KD, Mannstadt M, McMullen CP, Shonka DC Jr, Shin JJ, Singer MC, Slough CM, Stack BC Jr, Tearney G, Thomas G, Tolley N, Vidal-Fortuny J, Randolph GW. Emerging Imaging Technologies for Parathyroid Gland Identification and Vascular Assessment in Thyroid Surgery: A Review From the American Head and Neck Society Endocrine Surgery Section. JAMA Otolaryngol Head Neck Surg. 2023 Mar 1;149(3):253-260. doi: 10.1001/jamaoto.2022.4421. PMID 36633855
- [Background] Chernock RD, Jackson RS. Novel Cause of 'Black Thyroid': Intraoperative Use of Indocyanine Green. Endocr Pathol. 2017 Sep;28(3):244-246. doi: 10.1007/s12022-016-9458-z. PMID 27797004
- [Background] DeLong JC, Ward EP, Lwin TM, Brumund KT, Kelly KJ, Horgan S, Bouvet M. Indocyanine green fluorescence-guided parathyroidectomy for primary hyperparathyroidism. Surgery. 2018 Feb;163(2):388-392. doi: 10.1016/j.surg.2017.08.018. Epub 2017 Nov 10. PMID 29129358